CLINICAL TRIAL: NCT01176279
Title: Randomised Clinical Trial to Evaluate the Obtention of Blood Samples Through an Arterial Catheter to Monitor Glycose Levels
Brief Title: Arterial Catheter to Monitor Glycemia
Acronym: CAT-GLIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Hospitalari de Vic (Other)
Responsible Party: Mrs. Marta Raurell-Torredà, Vic Hospital Consortium - Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CGLIC-2007-03
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Critical Illness; Hyperglycemia
Keywords: Critical illness; Hyperglycemia; Catheters, Indwelling; Intensive care unit
MeSH Terms: conditions — Critical Illness; Hyperglycemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual and automated washing of the line (Active Comparator): Place in the radial artery the system of invasive monitoring of the blood pressure (BD DTXPlus ™). Insert in line a second 3-way stopcock above the one that has the BD DTXPlus ™; this second 3-way stopcock will be called proximal key. On the distal 3-way stopcock key (the one of TM BD DTXPlus ™), put the needless connector included in the kit to make the extractions of blood. Connect an arterial blood sampling syringe on the proximal 3-way stopcock key. With the assembled system, it is necessary to print a curve of invasive determination of the blood pressure.
  Interventions: Procedure: Manual and automated washing of the peripherical lines
- Automated washing of the line (Experimental): Place in the radial artery the system of invasive monitoring of the blood pressure (BD DTXPlus ™). Insert in line a second 3-way stopcock above the one that has the BD DTXPlus ™; this second 3-way stopcock will be called proximal key. On the distal 3-way stopcock key (the one of BD DTXPlus™), put the needless connector included in the kit to make the extractions of blood. On the proximal 3-way stopcock key put a second identical needless connector: in the intervention group the two 3-way stopcock keys have, each one, a needless connector. With the assembled system, it is necessary to print a curve of invasive determination of the blood pressure.
  Interventions: Procedure: Automated washing of the peripherical lines

INTERVENTIONS:
Procedure: Manual and automated washing of the peripherical lines — The extractions of the blood for the analysis of the glycaemia will be made puncturing the needless connector inserted in the distal 3-way stopcock key once an hour during 48 hours.
  Obtain 2cc of blood using the arterial blood sampling syringe connected to the proximal key. This volume of rejection is reserved in the syringe itself.
  In accordance with the current protocol of disinfection, the needless connector inserted on the distal key will be disinfected. With a disposable sterile syringe the needless connector is punctured and a minimum blood amount is obtained for the determination of the glycaemia.
  Once the sample has been obtained, the rejection volume reserved is returned to the bloodstream. This arterial blood sampling syringe is cleaned aspirating serum manually in order to wash the line.
  Additional line washing is made through the fast flow valve of the system BD DTXPlus ™.
  Arms: Manual and automated washing of the line
Procedure: Automated washing of the peripherical lines — The extractions of the blood for the analysis of the glycaemia will be made puncturing the needless connector inserted in the distal 3-way stopcock key once an hour during 48 hours.
  In accordance with the current protocol of disinfection, the two needless connectors inserted on the two 3-way stopcock keys will be disinfected.
  With a disposable sterile syringe the needless connector on proximal 3-way stopcock is punctured and 2cc of blood are aspirated. This volume of rejection is reserved in the syringe itself and it is not disconnected.
  With a second disposable sterile syringe the needless connector on distal 3-way stopcock key is punctured and a minimum blood amount is obtained for the determination of the glycaemia.
  Once the sample has been obtained, the rejection volume reserved in the disposable syringe connected to the proximal 3-way stopcock is returned to the bloodstream.
  Line washing will be made through the fast flow valve of the system BD DTXPlus ™.
  Arms: Automated washing of the line

SUMMARY:
The technique of blood samples extraction from the radial artery through an arterial catheter with a 3-way stopcock and automated washing with valve of fast flow is better than the one carried out through a fixed reusable arterial blood sample syringe and its manual washing because it shows a minor incidence of the complications originated from technical manipulation as infection, pseudo-aneurysm, ischemia or thrombosis of radial artery or obstruction of the catheter.

The purpose of this study is to evaluate the efficacy, in terms of adverse effects, of blood samples obtention using an arterial catheter with needless connector closed system or an arterial catheter with an arterial blood sample syringe.

Also a second purpose is to compare once a day (at the same time) the values of glycose blood levels between bedside glucometer determination of arterial catheter extraction and capillar puncture, and lab determination of glycose from venous puncture, in order to determinate fluctuation in glycose levels due to peripherical hypoperfusion or to vasoactive drugs received by these in-intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission in intensive care unit
* Insertion of a radial artery catheter for the invasive monitoring of haemodynamic pressure for a maximum of 5 days
* Need of insulin therapy by an intravenous continuous perfusion

Exclusion Criteria:

* Patients who do not accept to participate (or their relatives do not accept)
* Patients with a medical limitation of effort therapy
* Patients with FloTrac sensor from Edwards Lifesciences which does not allow to add a supplementary 3-way stopcock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Bacteremia episode originated from arterial catheter | At catheter's withdrawal (at seventh day of insertion or at any moment for any clinical reason)
  Catheter-related bloodstream infection as defined in Appendix A of "Guidelines for the Prevention of Intravascular Catheter-Related Infections". Centers for disease control and prevention (CDC) 2002 August 9: 51(RR10); 27.

SECONDARY OUTCOMES:
Local infection at cutaneous point of arterial catheter insertion | At catheter's withdrawal (at seventh day of insertion or at any moment for any clinical reason)
  Exit site infection as defined in Appendix A of "Guidelines for the Prevention of Intravascular Catheter-Related Infections". Centers for disease control and prevention (CDC) 2002 August 9: 51(RR10); 27.
Catheter colonization | At catheter's withdrawal (at seventh day of insertion or at any moment for any clinical reason)
  Localized catheter colonization as defined in Appendix A of "Guidelines for the Prevention of Intravascular Catheter-Related Infections". Centers for disease control and prevention (CDC) 2002 August 9: 51(RR10); 27.
Radial artery pseudo-aneurysm | Between 48 and 96 hours after catheter's withdrawal
  Diagnosed by the means of Doppler ultrasonography
Ischemia or thrombosis of radial artery | Between 48 and 96 hours after catheter's withdrawal
  Diagnosed by the means of Doppler ultrasonography
Arterial catheter obstruction | From the date of arterial catheter insertion to withdrawal at seventh day or at any moment for any clinical reason
  Blood sample obtention from arterial catheter is unavailable.
Glycose blood levels | During the two days of catheter manipulation

CONTACTS AND LOCATIONS:
Overall Officials: Marta Raurell-Torredà, Principal Investigator — Vic Hospital Consortium - Consorci Hospitalari de Vic
Locations (1):
- Vic Hospital Consortium - Consorci Hospitalari de Vic, Vic, Catalonia, Spain

REFERENCES:
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Kulkarni A, Saxena M, Price G, O'Leary MJ, Jacques T, Myburgh JA. Analysis of blood glucose measurements using capillary and arterial blood samples in intensive care patients. Intensive Care Med. 2005 Jan;31(1):142-5. doi: 10.1007/s00134-004-2500-5. Epub 2004 Nov 23. PMID 15565362
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] Lacara T, Domagtoy C, Lickliter D, Quattrocchi K, Snipes L, Kuszaj J, Prasnikar M. Comparison of point-of-care and laboratory glucose analysis in critically ill patients. Am J Crit Care. 2007 Jul;16(4):336-46; quiz 347. PMID 17595363
- [Background] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA. Guidelines for the prevention of intravascular catheter-related infections. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 Aug 9;51(RR-10):1-29. PMID 12233868
- [Result] Peruzzi WT, Noskin GA, Moen SG, Yungbluth M, Lichtenthal P, Shapiro BA. Microbial contamination of blood conservation devices during routine use in the critical care setting: results of a prospective, randomized trial. Crit Care Med. 1996 Jul;24(7):1157-62. doi: 10.1097/00003246-199607000-00015. PMID 8674328
- See also: Arterial Catheter to Monitor Glycemia — http://www.chv.cat